CLINICAL TRIAL: NCT02173509
Title: An Educational Intervention to Improve the Use of Antibiotics in Portuguese Health Professional: Cluster-randomized Trial
Brief Title: An Educational Intervention to Improve the Use of Antibiotics in Portuguese Health Professional
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Principal Investigator, Maria Teresa Herdeiro, Prof, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PTDC/SAU-ESA/105530/2008
Record Dates: First submitted 2014-06-17; First posted 2014-06-25 (Estimated); Results first posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2022-09

CONDITIONS: Antibiotics Misuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational multifaceted intervention (Experimental): Multidisciplinary and multifaceted educational intervention about antibiotic prescription and dispense, in physicians and pharmacists.
  Interventions: Other: Multidisciplinary and multifaceted educational intervention.
- Control (No Intervention): Physicians and pharmacists that not received the multidisciplinary and multifaceted educational intervention about antibiotic prescription and dispense.

INTERVENTIONS:
Other: Multidisciplinary and multifaceted educational intervention. — Outreach visits (40 minutes) which included a PowerPoint presentation and impress materials: poster; flyers; participation certificate and articles mentioned in the presentation. This outreach visit aimed to change the knowledge-attitudes previously identified in a previous study as being associated with poor prescribing of antibiotics in the case of physicians and propensity to dispense antibiotics without medical prescription in the case of pharmacists.
  Arms: Educational multifaceted intervention

SUMMARY:
This is a cluster randomised controlled trial covering all general practitioners working in the National Health System (SNS) and all pharmacists working in community pharmacies in the area covered by the Health Region Administration of Center (ARS-C) . A specific educative intervention, designed from gaps detected in knowledge and attitudes with respect to antibiotics and resistance, will be carried out on the intervention group. The control group will not receive any specific intervention.

Hypotheses:

1. The attitudes and knowledge towards antibiotics generate habits of prescription by physicians
2. The attitudes and knowledge towards to antibiotics generate propensity to dispense antibiotics without prescription by pharmacists
3. The identification of the attitudes, knowledge and factors that generate habits of inadequate prescription will allow the design of specific educative interventions to improve the use of antibiotics
4. The identification of the attitudes, knowledge and factors that generate propensity to dispense antibiotics without prescription will allow the design of specific educative interventions to antibiotic use
5. The interventions designed from gaps detected in knowledge and attitudes with respect to antibiotics and resistance will improve the prescription and dispensation of antibiotics by physicians and pharmacists, respectively.
6. The intervention will collaborate in the control of the bacterial resistance.

DETAILED DESCRIPTION:
The intervention will consist of group outreach visits (40 minutes), and will be targeted at changing the knowledge-attitudes previously found to be associated with poor prescribing of antibiotics in the case of physicians and propensity to dispense antibiotics without medical prescription in the case of pharmacists.. An observational cohort study of a sample of 1100 primary care physicians and 1200 community pharmacists will be carried out to identify knowledge-attitudes associated with inappropriate prescribing of antibiotics. The independent variables (knowledge-attitudes) will be assessed by a self-administered postal questionnaire and dependent variables are some quantity and quality indicators of the prescribing antibiotics, and consumption data.

ELIGIBILITY:
Inclusion Criteria:

* All general practitioners working during the period of the study in the National System of Health (SNS)
* All pharmacists working during the period study in the community pharmacies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2017-12 (Actual)

REFERENCES:
- [Derived] Teixeira Rodrigues A, Roque F, Pineiro-Lamas M, Falcao A, Figueiras A, Herdeiro MT. Effectiveness of an intervention to improve antibiotic-prescribing behaviour in primary care: a controlled, interrupted time-series study. J Antimicrob Chemother. 2019 Sep 1;74(9):2788-2796. doi: 10.1093/jac/dkz244. PMID 31257435
- [Derived] Roque F, Teixeira-Rodrigues A, Breitenfeld L, Pineiro-Lamas M, Figueiras A, Herdeiro MT. Decreasing antibiotic use through a joint intervention targeting physicians and pharmacists. Future Microbiol. 2016 Jul;11:877-86. doi: 10.2217/fmb-2016-0010. Epub 2016 Jul 14. PMID 27415585

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control group (n~ 791 GPs and n~888 pharmacists), not received the intervention.
- Intervention Group: The intervention group (n~ 309 GPs and n~312 pharmacists). Received the intervention (n~ 197 GPs and n~173 pharmacists)
Period: Overall Study
Arm/Group | Control Group | Intervention Group
Started | 1679 | 621
Completed | 1679 | 621
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The objective of the study is to evaluate the effectiveness of a joint educational intervention on overall antibiotic use, targeted at primary care physicians and community pharmacists.The sociodemographic data was not collected for this educational intervention study.We collected this data (age, sex) during the cross-sectional and cohort studies.
Groups:
- Intervention Group: Intervention group (n~ 309 GPs and n~312 pharmacists). Attended to the intervention, (n~ 197 GPs and n~173 pharmacists).
- Control Group: Intervention group (n~ 791 GPs and n~888 pharmacists).
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 621 | 1679 | 2300
Age, Categorical [Count of Participants; unit: Participants] — Population: Data not collected
Sex: Female, Male [Count of Participants; unit: Participants] — Data not collected. Population: data not collected
Region of Enrollment [Number; unit: participants]
  Portugal | 621 | 1679 | 2300

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Antibiotic Consumption at 18 Months, in Primary Care
Description: To quantify antibiotic drug consumption, we used monthly sales data sourced from IMS Health® and we used the quality indicators validated by Coenen S et al., (2007) to calculate monthly prescribing rates.
Time Frame: up to 18 months
Population: The analysis was performed with the intention to treat and the PID was assessed. These values correspond to the post-intervention period.
Measure: Mean (95% Confidence Interval); unit: PID-number of packages per 1000 inhabit
Groups:
- Control Group: Did not received in the multidisciplinary and multifaceted educational intervention about antibiotic prescription and dispense.
Arm/Group | Educational Multifaceted Intervention | Control Group
Number analyzed (Participants) | 621 | 1679
PID-number of packages per 1000 inhabit | 1.71 [1.65 to 1.77] | 2.01 [1.97 to 2.05]

2. Primary Outcome: Antibiotic Monthly Sales Data and Quality Indicators Monthly Prescribing Rates.
Description: antibiotic monthly sales data, obtained from IMS and quality indicators monthly prescribing rates, according to the ESAC indicators.
Time Frame: May 2012- September 2014
Measure: Mean (95% Confidence Interval); unit: PID-number of packages per 1000 inhabit
Groups:
- Control Group: Control group (n~ 791 GPs and n~ 888 pharmacists) Not attending to the intervention.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 621 | 1679
PID-number of packages per 1000 inhabit | 1.71 [1.65 to 1.77] | 2.01 [1.97 to 2.05]

ADVERSE EVENTS:
Description: The educational intervention, was an intervention to change behavior and knowledge of antibiotic use and not a clinical trial with medicines.
Groups:
- Control Group: The control group (n~791 GP and n~888 pharmacists) Not attending to the intervention.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes